CLINICAL TRIAL: NCT02974829
Title: A 5-Year Follow-up Study of Subjects Who Completed REALM-China Study
Brief Title: REALM China Extension Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463520
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Continuing with marketed anti-HBV or off-treatment in real-life setting
  Interventions: Other: follow-up

INTERVENTIONS:
Other: follow-up

SUMMARY:
The purpose of this study is to conduct an investigator initiated observational study to continue to follow up the China subset of study participants for another 5 years after they complete participation in the REALM Study

ELIGIBILITY:
Inclusion Criteria:

1. Patients completed REALM Study in China
2. Patients willing to sign the consent to continue anti-viral treatment or post-treatment follow up, and agree his/her legacy data and blood/liver histology samples collected in REALM Study may be used for the analyses planned for this new study.

Exclusion Criteria:

1. Patients who do not provide consent to participate in this study;
2. Patients are formally enrolled into any investigational drug clinical trial after the REALM study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-05; Primary Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Treatment patterns in Study AI463520 | year 5
Incidence rates of hepatitis B virus (HBV)-related clinical outcome events (COEs), such as non-hepatocellular carcinoma (HCC) HBV progression, HCC, and liver-related mortality, in Studies AI463080 and AI463520 combined, and in Study AI463520. | year 5

SECONDARY OUTCOMES:
Antiviral efficacy endpoints on anti-HBV treatment in Studies AI463080 and AI463520. | year 5
Multivariate logistic regression models evaluating the relationship between pre-treatment biomarkers and antiviral efficacy endpoints on anti-HBV treatment in Study | year 5
Multivariate logistic regression models evaluating the relationship between baseline liver stiffness measurement (LSM) and HBV-related COEs outcomes in Study AI463520. | year 5

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - People's Hospital of Beijing University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - GuangZhou No. 8 People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guiyang Medical College, Guiyang, Guizhou
  - People's hospital of Hainan Province, Haikou, Hainan
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Medical Science Research Institute of Henan Province, Zhengzhou, Henan
  - People's Hospital of Henan Province, Zhengzhou, Henan
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - No.81 Hospital of PLA, Nanjing, Jiangsu
  - The second hospital of nanjing, Nanjing, Jiangsu
  - Ningbo infectious disease hospital, Ningbo, Jiangsu
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - People's hospital of Jiangsu Province, Suzhou, Jiangsu
  - First Hospital of Jilin Unniversity, Changchun, Jilin
  - No.6 People's hospital of Dalian, Dalian, Liaoning
  - ShengJing Hospital of China Medical University, Shengyang, Liaoning
  - No.6 People's hospital of Shenyang, Shenyang, Liaoning
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Jinan infectious disease hospital, Jinan, Shandong
  - No.85 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital of SiChuan University, Chengdu, Sichuan
  - The first affiliated hospital of kunming medical college, Kunming, Yunnan
  - First Affiliated Hospital of Zhejing University, Hangzhou, Zhejiang
  - Hangzhou No.6 people's hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - First Affiliated Hospital of Beijing University, Beijing
  - You An Hospital, Beijing
  - Southwest Hospital Affiliated the Third Military Medical University, Chongqing
  - Changhai Hospital of the Second Military Medical University of Chinese PLA, Shanghai
  - Huashan hospital of fudan university, Shanghai
  - Renji Hospital of Shanghai Jiao Tong University, Shanghai
  - Shanghai jing 'an district central hospital, Shanghai
  - Shanghai No.5 People's Hospital, Shanghai
  - Shanghai Public Health Clinical Center, Shanghai
  - Zhongshan Hospital of Fudan University, Shanghai
  - No.3 people's hospital of shenzhen, Shenzhen
  - Tianjin infectious disease hospital, Tianjin
  - Tianjin third central hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided